CLINICAL TRIAL: NCT00136058
Title: Randomized Trial of Osteoporosis Intervention Strategies in Hip Fracture Patients
Brief Title: Trial of Osteoporosis Intervention Strategies in Hip Fracture Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Heritage Foundation for Medical Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Hipfracture1; AHFMR 200100791-2
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-12

CONDITIONS: Osteoporosis
Keywords: osteoporosis; hip fracture
MeSH Terms: conditions — Osteoporosis; Hip Fractures | interventions — Absorptiometry, Photon; Alendronate; Risedronic Acid

INTERVENTIONS:
Procedure: bone densitometry (DEXA)
Drug: alendronate or risedronate

SUMMARY:
The objective of this study is to determine if an intervention with a fracture manager to arrange bone densitometry after a hip fracture is more effective in diagnosing and treating osteoporosis when compared to "usual care". "Usual care" consists of no intervention to arrange bone mineral density (BMD) testing or therapy other than what normally occurs in the community. The investigators postulate that a fracture manager will be more effective in getting BMD done and in starting appropriate therapy.

DETAILED DESCRIPTION:
All hip fracture patients in the Edmonton area will be screened for eligibility (mini-mental status >20, not on active osteoporosis pharmacologic therapy). All patients will have informed consent obtained. Patients will be randomized to 2 groups:

* Group 1: Active intervention. The fracture manager will arrange for bone densitometry (DEXA) to be done 3-6 months after the fracture. If the patient meets standard criteria for osteoporosis, therapy with a bisphosphonate (alendronate or risedronate) will be instituted by the study physicians.
* Group 2: Usual care. Patients will receive basic information about calcium and vitamin D and osteoporosis and told to follow up with their family doctor. At 6 months, patients will be contacted to determine if they have had a BMD done or started on active (drug) osteoporosis therapy. If not, the fracture manager will arrange the BMD and if appropriate therapy will be started by the study physicians.

All patients will be followed for 1 year. The primary endpoints are the number of patients who get a BMD and the number who are started on active osteoporosis therapy.

ELIGIBILITY:
Inclusion Criteria:

* Ages 50 or over; males or females.
* Reside in the community or have access to bone densitometry
* Hip fracture
* Patient can consent or proxy consent available
* No contraindications to bisphosphonates

Exclusion Criteria:

* Patient refuses consent process
* Already receiving active drug therapy for osteoporosis other than calcium and vitamin D
* Dementia or delirium
* Pathological fracture
* Chronic corticosteroid therapy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2002-01; Study Completion 2006-04

PRIMARY OUTCOMES:
the number of patients who get a BMD and the number who are started on active osteoporosis therapy

CONTACTS AND LOCATIONS:
Overall Officials: Donald W Morrish, MD, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada